CLINICAL TRIAL: NCT02676674
Title: Vitamin D Levels in Subjects With Vitamin D Deficiency Following Topical Application of Three Doses of Vitamin D Ointment - A Proof of Concept Study
Brief Title: Vitamin D Levels Following Topical Application of Vitamin D Ointment
Acronym: VITD-001
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: University of Minnesota (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: 602M84081
Record Dates: First submitted 2016-02-03; First posted 2016-02-08 (Estimated); Last update posted 2019-11-01 (Actual); Status verified 2019-10

CONDITIONS: Vitamin D Deficiency
MeSH Terms: conditions — Vitamin D Deficiency | interventions — Cholecalciferol

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Dose 1 (Experimental): Three topical applications of 100,000 units for a total of 300,000 units of vitamin D3 in a newly formulated ointment will be applied to the upper arms over three weeks.
  Interventions: Drug: Dose 1
- Dose 2 (Experimental): Three topical applications of 300,000 units for a total of 900,000 units of vitamin D3 in a newly formulated ointment will be applied to the upper arms over three weeks.
  Interventions: Drug: Dose 2

INTERVENTIONS:
Drug: Dose 1 — Subjects with vitamin D deficiency will be given 100,000 units of topical vitamin D on days 0,7, and 14. Vitamin D levels will be checked on days 7, 14, and 21.
  Other Names: cholecalciferol; 25-OH Vitamin D
  Arms: Dose 1
Drug: Dose 2 — Subjects with vitamin D deficiency will be given 300,000 units of topical vitamin D on days 0,7, and 14. Vitamin D levels will be checked on days 7, 14, and 21.
  Other Names: cholecalciferol
  Arms: Dose 2

SUMMARY:
This is a pre-post open label trial to assess the change in Vitamin D blood levels following treatment with three doses of topical Vitamin D3 in subjects with existing Vitamin D deficiency.

DETAILED DESCRIPTION:
The proposed study investigates safety and efficacy of a new topical vitamin D3 compound. The purpose of this Phase 1 trial is to determine whether topical application makes Vitamin D bioavailable to the systemic circulation in sufficient quantities to treat hypovitaminosis D. The study will assess the change in serum 25-hydroxy (25-OH) vitamin D concentrations following 3 doses of 100,000 IU or 3 doses of 300,000 IU of topical vitamin D3 ointment in volunteers with vitamin D deficiency. Adults with serum 25-OH vitamin D concentrations of < 20 ng/ml will receive a total of 300,000 IU or 900,000 IU in divided doses of topical vitamin D once per week for three weeks. Two 0.75 ml applicators of ointment will be applied to each upper arm (50,000 IU or 150,000 IU per arm) by study staff. Blood will be drawn at baseline prior to the first dose (Day 0) and on Days 7, 14, and 21. Total serum 25-OH vitamin D will be assayed at each draw. Parathyroid hormone, a measure of clinical effects of low vitamin D levels, will be checked at baseline and on day 21. Serum albumin adjusted calcium levels will be checked with each draw to check for possible effects of too much vitamin D absorption. The study will determine whether the topical application of Vitamin D ointment is able to correct existing vitamin D deficiency.

ELIGIBILITY:
Inclusion Criteria:

1. Known vitamin D deficiency based on blood work obtained prior to study consent defined as serum 25-hydroxyvitamin D less than or equal to 20 ng/mL within 30 days prior to study entry.
2. Adult, age 18 to 85 years, male or female
3. If on oral vitamin D therapy, have been on a stable dose for the previous 90 days.

Exclusion Criteria:

1. History of chronic liver disease with elevated liver function tests, chronic kidney disease (stage 3 or greater, eGFR <60 mL/min), uncontrolled thyroid disease (elevated thyroid function tests), primary or secondary hyperparathyroidism, hypercalcemia, or multiple endocrine neoplasia.
2. Hypercalcemia defined as either elevated corrected serum calcium >10.2 mg/dL) measured within 3 months prior to study.
3. estimated glomerular filtration rate (eGFR) <60 mL/min within 3 months prior to study.
4. Active cancers
5. Women who are pregnant or breastfeeding.
6. Individuals who are unable to give informed consent
7. Individuals with psoriasis, active eczema or other skin disease, or who are currently receiving treatments or medications for skin disease.
8. Individuals who do not agree to refrain from using tanning beds for the duration of the study.
9. Individuals who do not agree to avoid submerging the ointment site in water for 8 hours after ointment application.

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2016-03; Primary Completion 2017-06-15 (Actual); Study Completion 2017-06-15 (Actual)

PRIMARY OUTCOMES:
Change in vitamin D | 4 weeks
  Two sample paired t test of pre and post total serum 25-OH vitamin D level

SECONDARY OUTCOMES:
Parathyroid hormone level | 4 weeks
  Two sample paired t test of pre and post total vitamin D level
Calcium level | 4 weeks
  Identification of any potential albumen adjusted hypercalcemia events
Skin irritation | 4 weeks
  Identification of any skin irritation events

CONTACTS AND LOCATIONS:
Overall Officials: Kevin A Peterson, MD, MPH, Principal Investigator — University of Minnesota
Locations (1):
- University of Minnesota Physicians - Phalen Village Clinic, Saint Paul, Minnesota, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Ginde AA, Liu MC, Camargo CA Jr. Demographic differences and trends of vitamin D insufficiency in the US population, 1988-2004. Arch Intern Med. 2009 Mar 23;169(6):626-32. doi: 10.1001/archinternmed.2008.604. PMID 19307527
- [Background] Tangpricha V, Pearce EN, Chen TC, Holick MF. Vitamin D insufficiency among free-living healthy young adults. Am J Med. 2002 Jun 1;112(8):659-62. doi: 10.1016/s0002-9343(02)01091-4. PMID 12034416

DOCUMENTS (2):
  • Study Protocol (2016-09-16): https://cdn.clinicaltrials.gov/large-docs/74/NCT02676674/Prot_000.pdf
  • Statistical Analysis Plan (2016-09-16): https://cdn.clinicaltrials.gov/large-docs/74/NCT02676674/SAP_001.pdf